CLINICAL TRIAL: NCT06275412
Title: Family mHealth Intervention to Improve Health Outcomes in Black Youth With Type 1 Diabetes
Brief Title: Family Intervention for Black Teens With Type 1 Diabetes
Acronym: 3Ms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Deborah Ellis, Ph.D., Professor of Family Medicine and Public Health Sciences Wayne State University School of Medicine, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-23-04-5675; 5R01MD018583-02 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes; Family Relations
Keywords: Type 1 Diabetes; mobile health; Family-based intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational Attention Control (EAC) + Standard Medical Care (Active Comparator)
  Interventions: Behavioral: Educational Attention Control (EAC)
- The 3Ms 2.0 Intervention + Standard Medical Care (Experimental)
  Interventions: Behavioral: The 3Ms 2.0 Intervention

INTERVENTIONS:
Behavioral: The 3Ms 2.0 Intervention — The 3Ms is a culturally tailored, mHealth intervention for primary caregivers of Black adolescents with T1D focused on promoting daily parental monitoring of adolescent diabetes care and delivered via an Internet platform, Computer Intervention Authoring System (CIAS). The intervention content is based on the Information-Motivation-Behavioral Skills (IMB) model. Caregivers randomized to The 3Ms receive 3 sessions. The caregiver is guided through each session by an interactive and emotive three-dimensional narrator that reads and speaks aloud. Additional intervention content includes brief videoclips to provide skills demonstrations of supportive parenting practices related to diabetes care and text message reminders. Each session is no more than 20 minutes in length. The intervention is delivered over a three-month window, with the two follow-up sessions available to be accessed by the caregiver at one-month intervals after completion of the initial session.
  Arms: The 3Ms 2.0 Intervention + Standard Medical Care
Behavioral: Educational Attention Control (EAC) — The EAC intervention consists of three sessions delivered in an mHealth format via the CIAS internet platform over three months, with access for a maximum of six months. EAC provides structured information on topics of interest to caregivers of adolescents with T1D such as travelling with diabetes, or emergency preparedness for persons with diabetes. All participants receive their standard medical care.
  Arms: Educational Attention Control (EAC) + Standard Medical Care

SUMMARY:
The purpose of this study is to conduct a multicenter, randomized effectiveness trial of The 3Ms 2.0 compared to an educational control condition for improving adolescent glycemic control and diabetes-related family relationships and reducing primary caregiver diabetes-related distress among Black adolescents with type 1 diabetes (T1D) and their primary caregivers. The proposed study would develop and test The 3Ms 2.0 adapted intervention when delivered using a mobile health approach (accessed via parents' cell phone). The intervention will also include new family intervention content (videoclips and text messages).

DETAILED DESCRIPTION:
The proposed study is a multi-center randomized controlled trial (RCT) examining the efficacy of The 3Ms 2.0 compared to an educational attention control condition (EAC) for improving adolescent glycemic control and diabetes-related family relationships and reducing primary caregiver diabetes-related distress among Black adolescents with type 1 diabetes (T1D) and their primary caregivers. A randomized, controlled, repeated measures design will be used. The study will use a sample of 216 Black adolescent-caregiver dyads. Participants will be recruited at two sites (University of Tennessee Health Sciences Center/ LeBonheur Children's Hospital and Children's National Hospital in Washington, DC). 108 families will be recruited at each of the two sites. Wayne State University (WSU) will function as the coordinating center for the trial and will be responsible for overseeing the adequacy of all aspects of trial management.

Participants will be randomly assigned in a 1:1 ratio to receive The 3Ms 2.0 plus standard medical care or EAC plus standard medical care. In the 3Ms 2.0 condition, primary caregivers will receive a brief (10-20 minute) 3 session computer-delivered intervention via their mobile device. The intervention is designed to increase parental daily supervision of adolescent diabetes management. In the control condition, primary caregivers will also receive 3 brief computer-delivered sessions where the content is information and facts about type 1 diabetes. The intervention content will be available to the primary caregiver during a six month window and can be completed at their convenience.

Data collection occurs in the families' home at baseline (T1), three months post-baseline (corresponding with the midpoint of the intervention window) (T2), six months post- baseline (corresponding with the end of the intervention window) (T3) and 12 months post-baseline (T4). Data completion can be completed via the Internet should families live outside a reasonable driving distance from the recruitment site. Data collection is completed by the adolescent and caregiver on a tablet computer and includes questionnaires to assess adolescent diabetes management, parental supervision of diabetes management, family relationships and youth quality of life. Blood will also be collected to measure HbA1c (mean blood glucose level). Medical record data will also be collected.

The data analyses will be intent-to-treat, meaning that all randomized participants are included regardless of the intervention dose received. Trial data will analyzed using the linear mixed effect model (LME) for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10 years, 0 months - 14 years, 11 months
* Diagnosed with Type 1 diabetes
* Diagnosed for at least 6 months
* Black
* Primary caregiver willing to participate
* Residence within 30 miles of a recruitment site
* Caregiver ownership of an Internet-enabled device (cell phone, laptop or desktop computer, tablet, etc)

Exclusion Criteria:

* Mental health conditions that might compromise data integrity (e.g., developmental delay, schizophrenia, psychosis, current suicidality, homicidality)
* Co-morbid medical condition resulting in atypical diabetes management (e.g., cystic fibrosis)
* Inability to speak or read English
* Child is in out-of-home placement

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | Baseline, 3 months, 6 months, and 12 months
  Hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Caregiver Diabetes Distress | Baseline, 3 months, 6 months, and 12 months
  Parent Problem Areas in Diabetes (P-PAID). The questionnaire's items are rated on a scale from 1 (not a problem) to 6 (serious problem). Higher scores reflect more diabetes distress
Diabetes-Specific Family Conflict | Baseline, 3 months, 6 months, and 12 months
  Diabetes Family Conflict Scale-Short Form (DFCS-SF). The questionnaire's items are rated on a scale from 1 (almost never) to 3 (almost always). Higher scores reflect more family conflict
Diabetes-Specific Parental Monitoring | Baseline, 3 months, 6 months and 12 months
  Parental Monitoring of Diabetes Care-Revised (PMDC-R). The questionnaire's items are rated from 1 to 5, with higher scores reflecting higher parental monitoring
Diabetes-Specific Family Support | Baseline, 3 months, 6 months and 12 months
  Diabetes Social Support Questionnaire-Family (DSSQ-Family). Items reflecting frequency of support are rated from 0 (never) to 5 (at least once a day). Items reflecting helpfulness of support are rated from 0(not at all) to 2 (very). Higher scores reflect more frequent family support and more helpful family support

OTHER OUTCOMES:
Illness Management | Baseline, 3 months, 6 months, and 12 months
  Diabetes Management Scale (DMS). The questionnaire's items are rated from 0 to 100. Higher scores reflect higher levels of diabetes care completion
Intervention Satisfaction | 6 months
  Exit interviews will be conducted to obtain caregiver perspectives regarding satisfaction with intervention content, delivery mode and dose using semi-structured interview guides.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Ellis, Ph.D., Principal Investigator — Wayne State University
Locations (4):
- United States (4):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Wayne Pediatrics, Detroit, Michigan
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - University of Tennessee Health Science Center-Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Identifiers will be removed from the data prior to any release of the dataset. The final data set will include data obtained from medical records, data obtained directly from participants on diabetes health status, behavioral data, and intervention data. Participants in the trial will be recruited through two children's hospitals. Even though the final dataset will not contain identifiers, given the relatively small sample size and focus on Black youth, there remains the possibility of deductive identification of subjects with unusual characteristics (i.e. high number hospital admissions).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2029
Access Criteria: Given the sensitive nature of the health data contained in the data set, as well as the participation of children, the data and associated documentation will be available to users under a specific data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate technology; and (3) a commitment to destroying the data after analyses are completed.